CLINICAL TRIAL: NCT02598154
Title: Evaluation of the Metrological Characteristics of the Inertial Unit FOX HiKoB© in Comparison With the Reference System for the Adaptive Trigger System "Functional Electrical Stimulation" of Foot Elevators in Hemiplegic Post-stroke Patients
Brief Title: Metrological Characteristics of the Inertial Unit "FOX HiKoB©" in Comparison With the Reference System for the Adaptive Trigger System "Functional Electrical Stimulation" of Foot Elevators in Hemiplegic Post-stroke Patients
Acronym: MASEA 2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/JF-01; 2015-A00572-47 (Other: ANSM)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: The study population consists of patients whose age is between 20 and 75 years and who experienced a supra-tentorial ischemic or hemorrhagic stroke. The study covers inpatients or patients consultating in the neurological rehabilitation service (NHS) at the Grau du Roi Medical Center, Nîmes University Hospital.

SUMMARY:
The main objective of this study is to evaluate the metrological characteristics of the data processing algorithms from inertial sensors (FOX © HiKoB) for the reconstruction of movement relative to the reference system (VICON) for measurement of dorsiflexion at the beginning of a step and in the middle of the oscillating phase.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

1. / - to assess the metrological characteristics of the data from inertial sensors (FOX © HiKoB) for the reconstruction of the movement in comparison with reference systems (GaitRite or Zebris systems, VICON) in terms of:

   A. Ability to determine the walking speed, stride length, the acceleration of plantar flexion at the beginning of the weight-bearing phase B. Ability to objectify performance reduction during a 6 minute test. C. Ability to identify different types of movement: simple walking, turn, obstacle clearance, staircase.
2. / - to analyze the EMG signal upon voluntary dorsiflexion of the foot of the paretic side from a sitting position before and after a fatigue test (objective D)

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Stroke, ischemic or hemorrhagic, supra-tentorial, regardless of the post-stroke period
* The patient can walk 10m without human help, with or without a cane and has a foot elevator deficit requiring the use of technical assistance or causing a walking defect

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient or his/her representative refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant or breastfeeding
* The patient has cognitive impairment
* Presence of permanent plantar flexion of the ankle joint with ankle dorsiflexion, knee straight, lower than 0°.
* Uncontrolled epilepsy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients whose age is between 20 and 75 years and who experienced a supra-tentorial ischemic or hemorrhagic stroke. The study covers inpatients or patients consultating in the neurological rehabilitation service (NHS) at the Grau du Roi Medical Center, Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Dorsiflexion (°) at the beginning of a step | Day 0
Dorsiflexion (°) in the middle of the oscillating phase | Day 0

SECONDARY OUTCOMES:
Walking speed | Day 0
Stride length | Day 0
Maximal angular speed at the ankle between the moment when the heel touches the ground and the moment where the foot is flat (°/s) | Day 0
6 minute walking test: average dorsiflexion ankle measured between 15 seconds and 30 seconds | Day 0
6 minute walking test: average dorsiflexion ankle measured between 30 seconds and 5 min 5 min 45 seconds | Day 0
Detection of obstables: yes/no | Day 0
EMG signal (%) during voluntary dorsiflexion of the foot of the paretic side in a sitting position before and after fatigue test | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Froger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Cristine Azevedo Coste, Study Director — DEMAR INRIA / LIRMM, 161 rue Ada, 30392 Montpellier Cedex 5
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Sijobert B, Feuvrier F, Froger J, Guiraud D, Coste CA. A sensor fusion approach for inertial sensors based 3D kinematics and pathological gait assessments: toward an adaptive control of stimulation in post-stroke subjects. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:3497-3500. doi: 10.1109/EMBC.2018.8512985. PMID 30441133